CLINICAL TRIAL: NCT03050177
Title: Single-dose, Open-label, Randomized, 2-way Crossover Bioequivalence Study of Gefitinib Tablets Under Fed Conditions in Chinese Healthy Male Subjects
Brief Title: Bioequivalence Study of Gefitinib Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hunan Kelun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: KL031-BE-02
Record Dates: First submitted 2017-01-21; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Bioequivalence Study
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefitinib Tablet 250mg of Hunan Kelun (Experimental): During the study session, healthy subjects were orally administered a single dose of Gefitinib Tablet 250mg of Hunan Kelun under fed conditions.
  Interventions: Drug: Gefitinib Tablet 250mg of Hunan Kelun; Drug: Iressa® Tablet 250mg of AZN
- Iressa® Tablet 250mg of AZN (Active Comparator): During the study session, healthy subjects were orally administered a single dose of Iressa® Tablet 250mg of AZN under fed conditions.
  Interventions: Drug: Gefitinib Tablet 250mg of Hunan Kelun; Drug: Iressa® Tablet 250mg of AZN

INTERVENTIONS:
Drug: Gefitinib Tablet 250mg of Hunan Kelun — Single dose of Gefitinib Tablet 250mg of Hunan Kelun was administered under fed conditions after a 10-hour overnight fast.
  Other Names: A031
Drug: Iressa® Tablet 250mg of AZN — Single dose of Iressa® Tablet 250mg of AZN was administered under fed conditions after a 10-hour overnight fast.
  Other Names: Iressa®

SUMMARY:
The study design is an Open-Label，Randomized, Single-Dose, 2-way Crossover Bioequivalence Study. During each session, the subjects will be administered a single dose of 250mg Gefitinib Tablet (one Gefitinib Tablet 250mg of Hunan Kelun or one Iressa® Tablet 250mg of AstraZeneca) under fed conditions.

DETAILED DESCRIPTION:
An Open-Label，Randomized, Single-Dose, 2-way Crossover Bioequivalence Study . During each session, the subjects were randomly assigned in a 1:1 ratio to receive a single 250-mg dose of either the test formulation(Hunam Kelun) or the reference formulation(Iressa® Astrazeneca), and vice versa, with a 21-day washout period between administration periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects.
2. At least 18 years of age .
3. Weight at least 50kg and body mass index between 19 and 26 kg/m2.
4. Informed consent and voluntary to sign a written informed consent.
5. Can communicate with researchers and complete the study in accordance with the provisions of the research.

Exclusion Criteria:

1. Abnormal diagnostic findings, and clinical significances determined by researchers (physical examination,vital sign, ECG,X-ray,blood routine examination, urine routine examination,blood biochemical examination and coagulation test).
2. Having functional gastrointestinal disease or inadequate secretion of gastric acid or is treated for a acid suppression. Which including gastro upset, dyspepsia, gastritis, gastric ulcer, duodenal ulcer, gastric secrete melanoma, etc.
3. Taking drugs that alter the environment of the gastrointestinal，especially alter the gastrointestinal pH，within 30 days before the first dose. Such as， Proton pump inhibitors：thiophene, omeprazole, lansoprazole, esomeprazole, etc .and H2 antagonist ranitidine：cimetidine, famotidine, etc .and antacids hydrogen carbonate Sodium, magnesium oxide, aluminum hydroxide, magnesium trisilicate, etc .and gastric mucosal protective agent：sucralfate，and so on.
4. Not comply with a unified diet( such as standard meal) or has swallowing difficulties.
5. Allergic to any ingredient or excipients of the study drug.
6. History of gastrointestinal disorders and severe liver and kidney diseases ，which affect the absorption or metabolism of drugs so far.
7. History of ocular surface damaging diseases (such as corneal perforation, ulcers, etc.).
8. History of serious blood diseases.
9. With skin, cardiovascular, liver, kidney, digestive, neurological, psychiatric, metabolic disorders, or any other disease that can interfere with the results of the trial.
10. History of long-term excessive drinking (more than 8 cups a day, 1 cup = 250 mL) of tea, coffee or caffeinated beverages，or 48 hours before the first dose intake of any food or drink containing caffeine (such as coffee, tea, chocolate, etc.).
11. Ingested any drinks or foods that are rich in xanthine and grapefruit or affect the drug absorption, distribution, metabolism and excretion.
12. A positive result in breath alcohol test or previous alcohol abuse (ie, men drink more than 28 standard units a week [1 standard unit defined as containing 14 grams of alcohol, such as would be found in a standard shot of hard liquor, a 12-ounce bottle of beer, or a 5-ounce glass of wine] Or regular drinking(more than 14 standard units of alcohol per week) within 6 months before the trial.
13. Daily intake of more than 3 cigarettes from 3 months before the study to 48 hours before the first dose or intake of tobacco or any type of tobacco product within 48 hours before the first dose.
14. Taking drugs that interact with gefitinib （such as CYP3A4 inhibitors： itraconazole, ketoconazole, clotrimazole, Ritonovir, etc .and CYP3A4/5 inducers：rifampicin, carbamazepine, phenobarbital, phenytoin, dexamethasone, etc .and CYP2D6 inhibitors：Fluoxetine, paroxetine , etc .） within 30 days before the first dose. And use of any prescription drugs, non-prescription drugs, Chinese herbal medicine, health products within 14 days before the first dose.
15. Volunteer in any other clinical drug study or taking any clinical trial drug within 3 months prior to this study.
16. Blood donation or lost more than 450mL blood within 3 months prior to the study，or has a plan to donate blood or blood components within the study period or within 3 months after the end of study.
17. Suffering from a serious illness or having undergone major surgical procedures within 1 years before the firs dose.
18. Abnormal blood coagulation, or having a known tendency of severe bleeding..
19. A positive result in drug test or existing drug abuse (eg, morphine, marijuana, methamphetamine, dimethylene bisoxamine amphetamines, ketamine, etc.) within 1 year prior to the trial.
20. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test.
21. Having fertility planning or reluctant to take appropriate contraceptive during the study or within 6 months after the study.
22. Other unfavorable factors diagnosed by investigators.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter：Cmax | before drug delivery through 216 hours after dosing
  Peak Plasma Concentration (Cmax)
Pharmacokinetic parameter：AUC | before drug delivery through 216 hours after dosing
  Area under the plasma concentration versus time curve (AUC)

IPD SHARING:
Plan to Share IPD: No